CLINICAL TRIAL: NCT01044589
Title: Comparison of the Efficacy of a Biological Implant to Reinforce Overlapping Sphincter Repair Versus Overlapping Sphincter Repair Alone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to low enrollment
Sponsor: Massarat Zutshi (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Massarat Zutshi, Staff, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-008
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Fecal Incontinence; Anal Incontinence
MeSH Terms: conditions — Fecal Incontinence; Encopresis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Biodesign Tissue Repair Graft (Experimental): Biodesign Tissue Repair Graft
  Interventions: Device: Biodesign Tissue Repair Graft; Other: Overlapping Sphincter Repair
- Overlapping Sphincter Repair (Active Comparator): Control
  Interventions: Other: Overlapping Sphincter Repair

INTERVENTIONS:
Device: Biodesign Tissue Repair Graft — Biodesign Tissue Repair Graft reinforcement
  Arms: Biodesign Tissue Repair Graft
Other: Overlapping Sphincter Repair — Overlapping Sphincter Repair Alone

SUMMARY:
The aim of this study is to compare the efficacy of Biodesign™ Surgisis® Tissue Graft to reinforce an overlapping sphincter repair versus the standard overlapping sphincter repair in controlling episodes of incontinence in patients who have fecal incontinence and a defect in the anal sphincter.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 years or older
* fecal incontinence due to an anterior defect in the external anal sphincter or both external and internal anal sphincter muscles
* Fecal incontinence severity score of 10 or more
* Fecal incontinence episodes of 4 or more over a 2 week period

Exclusion Criteria:

* History of diabetes
* History of allergy to porcine derivatives
* History of infection in the anal area (abscess, fistula)
* History of inflammatory bowel disease
* History of hidradenitis suppurativa
* History of immunosuppression
* History of HIV positivity
* History of radiation to the study site within the last 12 months
* Patients who cannot travel to keep follow up appointments
* Patients who are prisoners
* Patients who are mentally handicapped
* Patients who are pregnant or plan to become pregnant during the study period, or who are currently breastfeeding
* Patients with significant posterior pelvic organ prolapse and who would be candidates for concomitant treatment.
* Patients with a FIQL baseline score of ≤ 4
* Patients participating in another clinical trial for the same indication
* Patients unwilling to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massarat Zutshi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overlapping Sphincter Repair | Biodesign Tissue Repair Graft
Started | 6 | 7
Completed | 3 | 2
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Overlapping Sphincter Repair | Biodesign Tissue Repair Graft | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting a Decrease in Incontinence Episodes Per Week
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overlapping Sphincter Repair | Biodesign Tissue Repair Graft
Number analyzed (Participants) | 3 | 3
Participants | 2 | 2

2. Secondary Outcome: Number of Participants Reporting a Decrease in Incontinence Episodes Per Week
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overlapping Sphincter Repair | Biodesign Tissue Repair Graft
Number analyzed (Participants) | 5 | 3
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Overlapping Sphincter Repair | Biodesign Tissue Repair Graft
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overlapping Sphincter Repair (N=6) | Biodesign Tissue Repair Graft (N=7)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No